CLINICAL TRIAL: NCT06871865
Title: The Effects of Oculomotor Training on Pain, Cervical Range of Motion, Joint Position Sense, Endurance, and Balance in Individuals With Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Eda AKBAŞ, Associate Professor, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BEUN-AKBAS-2
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-03

CONDITIONS: Mechanical Neck Pain
Keywords: Mechanical neck pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): This group will be given a home program including isometric neck strengthening exercises, neck stretching exercises and posture exercises during the 6-week treatment period, and the control group will be given an additional oculomotor exercise program.
  Interventions: Other: Oculomotor Exercises; Other: Posture Exercises; Other: Neck Stretching and Strengthing Exercises
- Control Group (Active Comparator): This group will be given a home program including isometric neck strengthening exercises, neck stretching exercises and posture exercises during the 6-week treatment period.
  Interventions: Other: Posture Exercises; Other: Neck Stretching and Strengthing Exercises

INTERVENTIONS:
Other: Oculomotor Exercises — Oculomotor exercises are designed to improve eye movement control, coordination, and visual tracking.
  Arms: Intervention Group
Other: Posture Exercises — Postural exercises help strengthen core muscles, improve alignment, and enhance stability. They are essential for maintaining proper posture, preventing pain, and reducing the risk of musculoskeletal imbalances.
Other: Neck Stretching and Strengthing Exercises — Neck stretching and strengthening exercises help improve flexibility, reduce stiffness, and enhance muscle support for the cervical spine. They are beneficial for relieving neck pain, improving posture, and preventing injuries.

SUMMARY:
The aim of this study was to investigate the effects of oculomotor training on pain, cervical range of motion, joint position sense, endurance and balance in individuals with mechanical neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mechanical neck pain
* Neck pain lasting longer than 3 weeks
* Individuals aged 18-50 years
* Score of 5 or higher on the Neck Disability Index

Exclusion Criteria:

* Having received physical therapy in the last 6 months
* Presence of congenital anomaly on cervical radiography
* Neurological deficit detected in physical examination
* Diagnosis of vertebrobasilar artery insufficiency
* Diagnosis of vestibular disease
* Presence of a rheumatic disease
* Presence of structural scoliosis
* History of spinal surgery
* Pregnancy
* Malignancy
* Eye disease/strabismus other than refractive errors
* Active use of anti-inflammatory medication
* Any mental condition that may prevent adherence to exercises

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | From enrollment to the end of treatment at 6 weeks

SECONDARY OUTCOMES:
Neck Disability Index | From enrollment to the end of treatment at 6 weeks
Craniovertebral Angle | From enrollment to the end of treatment at 6 weeks
Cervical ROM | From enrollment to the end of treatment at 6 weeks
  Flexion, extension, lert-right rotation, left-right lateral flexion will be measured.
Craniocervical Flexion Test | From enrollment to the end of treatment at 6 weeks
  Endurance of the deep cervical flexor muscles will be measured.
Y Balance Test | From enrollment to the end of treatment at 6 weeks
  Y Bavlance Test will be applied to test the ability to reach of upper extremity.
Beck Depression Inventory | From enrollment to the end of treatment at 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Zonguldak Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided